CLINICAL TRIAL: NCT06318247
Title: Using Xenograft Combined With Barrier Membrane to Improve the Formation of Deep Periodontal Pockets in the Distal of the Mandibular Second Molar After the Extraction of the Third Molar
Brief Title: Using Xenograft Combined With Barrier Membrane to Improve the Formation of Deep Periodontal Pockets
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-134(R)
Record Dates: First submitted 2023-08-27; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Periodontal Pocket; Periodontal Bone Loss; Impacted Third Molar Tooth
MeSH Terms: conditions — Periodontal Pocket; Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Tooth extraction of third molars
  Interventions: Procedure: site preservation
- GBR group (Experimental): Tooth extraction of third molars with site preservation using bio-oss (0.5g, Small granule) and bio-guide (25*25mm size). The bone graft material used in the surgical procedure was provided by Geistlich Pharma AG.
  Interventions: Procedure: site preservation

INTERVENTIONS:
Procedure: site preservation — Tooth extraction of third molars with site preservation using bio-oss (0.5g, Small granule) and bio-guide (25*25mm size). The bone graft material used in the surgical procedure was provided by Geistlich Pharma AG.

SUMMARY:
To evaluate the clinical effect of site preservation after third molars extraction by using tooth extraction of third molars with site preservation using bio-oss and bio-guide in preventing the formation of deep periodontal pockets in the distal of second molars.

DETAILED DESCRIPTION:
The mandibular third molar is the last tooth to erupt in the dentition, and due to the insufficient eruption position, it can lead to different degrees of impact. During the eruption of impacted tooth, the crown may be partially or completely covered by the gingival flap. A deep blind pocket is formed between the gingival flap and the tooth crown, and food and bacteria are easily impinged in the blind pocket. Under the influence of oral environment and dental plaque, the presence of blind pockets can lead to the loss of periodontal attachment and the absorption of alveolar bone, thus affecting the distal periodontal status of adjacent molars.

Organic bone xenograft material composed of absorbable organic bovine hydroxyapatite is one of the commonly used transplantation materials for repairing bone defects. The application effect of allogeneic bone materials in periodontal therapy has been recognized by many experts and scholars. Guided bone regeneration (GBR), as a conventional periodontal bone graft, has achieved good results in periodontal tissue regeneration. Aljuboori et al. found that when the third molar was removed and GBR was performed at the same time, the depth of distal periodontal pocket probing of the adjacent second molar was significantly reduced in the re-examination 6 months after surgery.

Hence, this study intends to use xenograft combined with barrier membrane to improve the formation of distal periodontal pocket of the second molars after third molars extraction.

ELIGIBILITY:
Inclusion Criteria:

* 26-45 years old
* Completely or partially impacted mandibular third molar
* No evidence of acute inflammation
* In good physical status and oral health
* Regular attendance at control visits

Exclusion Criteria:

* pregnancy or lactation
* Aggregate systemic pathologies such as diabetes, thyroid disorders, bone metabolism diseases, among others
* Patients taking calcium, bisphosphonates, glucocorticoids, or other drugs that can interfere with bone metabolism
* Patients with uncontrolled periodontal conditions, endodontic conditions and other oral disorders
* Heavy smoke (10 cigarettes/day or more)
* The second molar has no contact with the third molar, or the third molar crown has alveolar bone

Ages: 26 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depths (PPD) | postoperative 14 days, 3 6 and 12 months
  The depth of the periodontal pocket is examined with a periodontal probe. Probing pocket depths (PPD) measured in millimeters at six sites: disto-vestibular (DV), centro-vestibular (CV), mesio-vestibular (MV), disto-lingual (DL), centro-lingual(CL), mesio-lingual (ML) in postoperative 14days, 3, 6 and 12 months. The distal measurements are the primary outcomes. The higher the value, the worse the periodontal condition.
Distal bone wall defect (DBWD) | postoperative 14 days, 3 6 and 12 months
  The height of distal bone wall defect of the second mandibular molar is measured by cone-beam CT.
Clinical attachment lose (CAL) | postoperative 14 days, 3 6 and 12 months
  clinical attachment lose (CAL) were measured in millimeters at six sites: disto-vestibular (DV), centro-vestibular (CV), mesio-vestibular (MV), disto-lingual (DL), centro-lingual(CL), mesio-lingual (ML). The distal measurements are the primary outcomes.
Bleeding on probing (BOP) | postoperative 14 days, 3 6 and 12 months
  Periodontal probing for bleeding can determine whether the gingiva is in a state of inflammation or whether periodontal disease is in an active phase.

SECONDARY OUTCOMES:
Pain score | pre-operation, postoperative 14 days, 3 6 and 12 months
  Visual Analog Score for pain
Patient satisfaction | pre-operation, postoperative 14 days, 3 6 and 12 months
  Physicians Global Assessment to measure quality of life
Gingival index (GI) | pre-operation, postoperative 14 days, 3 6 and 12 months
  The higher the index, the worse the periodontal condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Stomatology Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China